CLINICAL TRIAL: NCT02230722
Title: Improving Opioid Safety in Veterans Using Collaborative Care and Decision Support
Acronym: OPTI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Karen Seal, Principal Investigator, San Francisco Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-11892; R34AT008319-01 (NIH)
Record Dates: First submitted 2014-08-25; First posted 2014-09-03 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Chronic Pain
Keywords: opioids; chronic pain; collaborative care
MeSH Terms: conditions — Chronic Pain | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Control (Active Comparator): The neutral 10-15 minute visit with the Care Manager will consist of a brief review of ATHENA-OT safety education and the patient's Pain Care Plan. The CM will answer patient questions, but will avoid using Motivational Interviewing communication. The Care Manager will review upcoming telephone check-in and assessment sessions.
  Interventions: Behavioral: Attention Control
- Collaborative Care (Experimental): Collaborative Care intervention in which one of two Care Managers delivering both interventions will assist primary care providers (PCPs) by using Motivational Interviewing to communicate computer-based ATHENA-OT (opioid therapy) decision support guidelines to veterans with chronic pain.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing
  Arms: Collaborative Care
Behavioral: Attention Control
  Arms: Attention Control

SUMMARY:
The investigators propose to develop a novel intervention that targets the system (Collaborative Care), PCP (computerized decision support for opioid therapy) and veteran (CM-delivered MI) to reduce problematic prescription opioid use and encourage non-opioid pain management alternatives.

DETAILED DESCRIPTION:
The investigators will develop and test the acceptability, feasibility, and preliminary efficacy of a Collaborative Care intervention in which one of two Care Managers delivering both interventions will assist primary care providers (PCPs) by using Motivational Interviewing to communicate computer-based ATHENA-OT (opioid therapy) decision support guidelines to veterans with chronic pain. Specifically, after honing the intervention, the investigators will conduct a pilot randomized controlled trial of Collaborative Care/Motivational Interviewing in 100 veterans (ages 18 and older) with chronic pain in primary care who are prescribed opioid pain medications and exhibit at least one "high-risk" opioid use behavior (e.g. obtaining early opioid refills, etc.). Using ATHENA-OT decision support, PCPs will make guideline-concordant recommendations to all enrolled study patients and initiate a Pain Care Plan. Veterans randomized to Collaborative Care, will have one MI session with their assigned study Care Manager followed by 3 Care Manager-delivered telephone MI/monitoring sessions; patients randomized to the Attention Control arm will have one brief session with their assigned Care Manager, followed by 3 Care Manager-delivered neutral telephone sessions

ELIGIBILITY:
Inclusion Criteria:

* Current Male or Female patient at San Francisco VA Medical Center or affiliated VA clinics
* Must be older than 18 years
* Chronic musculoskeletal pain of at least 6 months duration and
* Prescribed one or more opioid pain medication for more than three months and
* Evidence of being a high-risk opioid user as determined by PI, electronic medical record, and study measures

Exclusion Criteria:

* Non-English speakers
* Plans to relocate within 6 months; not able to come to San Francisco VA Medical Center for three in-person visits
* Cancer or other terminal illness involving palliative care with opioid medications
* Serious or untreated mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility, acceptability, and usability of augmenting ATHENA-OT decision support with a Collaborative Care intervention. | 20 weeks post baseline
  * PCPs and the CM in the Collaborative Care arm will report greater self-efficacy in communicating ATHENA-OT pain management recommendations and in developing a Pain Care Plan with chronic pain patients
  * The CM will conduct MI communication with high fidelity.
  * Veterans in the Collaborative Care arm will report greater satisfaction with pain-related care.

SECONDARY OUTCOMES:
To preliminarily evaluate the efficacy of ATHENA-OT decision support plus Collaborative Care (CC) to improve prescription opioid safety and adherence to non-opioid pain management alternatives among primary care patients. | 20 weeks post baseline
  Compared to ATHENA-OT plus Attention Control:
  H2.a. Veterans randomized to Collaborative Care (CC) will be more likely to achieve a decrease in opioid risk behavior that is sustained during an 8-week post-intervention period of no contact.
  H2.b. Veterans randomized to CC are more likely to initiate and sustain ≥ 1 non-opioid strategies.
  H2.c. Veterans randomized to CC are more likely to report sustained improvements in pain disability.
  H2.d. Substance use disorders and treatment will moderate CC efficacy; Care Manager MI-consistent communication in the CC arm will correlate with reduced opioid risk behavior in veterans.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Seal, MD, MPH, Principal Investigator — SFVAMC
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Okie S. A flood of opioids, a rising tide of deaths. N Engl J Med. 2010 Nov 18;363(21):1981-5. doi: 10.1056/NEJMp1011512. No abstract available. PMID 21083382
- [Background] Paulozzi LJ, Kilbourne EM, Desai HA. Prescription drug monitoring programs and death rates from drug overdose. Pain Med. 2011 May;12(5):747-54. doi: 10.1111/j.1526-4637.2011.01062.x. Epub 2011 Feb 18. PMID 21332934
- [Background] Boudreau D, Von Korff M, Rutter CM, Saunders K, Ray GT, Sullivan MD, Campbell CI, Merrill JO, Silverberg MJ, Banta-Green C, Weisner C. Trends in long-term opioid therapy for chronic non-cancer pain. Pharmacoepidemiol Drug Saf. 2009 Dec;18(12):1166-75. doi: 10.1002/pds.1833. PMID 19718704
- [Background] Paulozzi LJ; Centers for Disease Control and Prevention (CDC). Drug-induced deaths - United States, 2003-2007. MMWR Suppl. 2011 Jan 14;60(1):60-1. No abstract available. PMID 21430623
- [Background] Seal KH, Shi Y, Cohen G, Cohen BE, Maguen S, Krebs EE, Neylan TC. Association of mental health disorders with prescription opioids and high-risk opioid use in US veterans of Iraq and Afghanistan. JAMA. 2012 Mar 7;307(9):940-7. doi: 10.1001/jama.2012.234. PMID 22396516
- See also: Veterans Return Home Research Group — http://vetsreturnhome.com/index.html